CLINICAL TRIAL: NCT02410070
Title: A Comparison of Minimal Approach With Conventional Approach for Distal Radial Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1011126
Record Dates: First submitted 2015-03-18; First posted 2015-04-07 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Closed Frykman Type II Fracture of Right Radial Head
Keywords: Distal radial fracture; pronator quadratus; mini-approach; volar plating; open reduction and internal fixation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Though Volar Minimal Incision (Experimental): Patients in group A were treated through a small Incision.
  Interventions: Procedure: Incision
- Though Convectional Incision (Active Comparator): Patients in group B were treated through the conventional Incision
  Interventions: Procedure: Incision

INTERVENTIONS:
Procedure: Incision — The objective of this report is to compare a minimal invasive approach with the conventional flexor carpi radialis approach for volar plating of distal radial fractures.

SUMMARY:
The objective of this study is to compare a minimal invasive approach with the conventional flexor carpi radialis approach for volar plating of distal radial fractures.

DETAILED DESCRIPTION:
The objective of this study is to compare a minimal invasive approach with the conventional flexor carpi radialis approach for volar plating of distal radial fractures.

From January 2011 to September 2012, 157 patients with distal radial fractures were allocated into group A (n=83) and B (n=74). Patients in group A were treated through a 1.5 to 2-cm long incision, and patients in group B were treated through the conventional flexor carpi radialis approach. All fractures were fixed with volar plates. Patients were assessed range of motion of the wrist, grip strength of the hand, and pronation strength of the wrist. Results were analyzed with the Statistical Package for Social Sciences 13.0. A P < 0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Fernandez type II-IV radial fractures.

Exclusion Criteria:

* Fernandez type I radial fracture.
* Fernandez type V radial fracture.
* Open radial fractures.
* Surgery using K-wires or screws alone.
* The use of external fixators.
* multiple fractures, pathological fracture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
range of motion of the wrist | 2 years
  measurement of range of motion of the wrist with a goniometer, at 2 years follow-up.

SECONDARY OUTCOMES:
grip strength of the hand | 2 years
  Assessment of grip strength of the hand using a Baseline hydraulic hand dynamometer, at 2 years follow-up.
pronation strength of the forearm | 2 years
  Isometric testing of pronation torque, McConkey method at 5 positions of rotation (90° of supination, 45° of supination, neutral, 45° of pronation, and 80° of pronation) , at 2 years follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Study Chair — The Second Hospital of Qinhunangdao

REFERENCES:
- [Result] Skouras E, Hosseini Y, Berger V, Wegmann K, Koslowsky TC. Operative treatment and outcome of unstable distal radial fractures using a palmar T-miniplate at a non-specialized institution. Strategies Trauma Limb Reconstr. 2013 Nov;8(3):155-60. doi: 10.1007/s11751-013-0170-y. Epub 2013 Aug 6. PMID 23918414
- [Result] Protopsaltis TS, Ruch DS. Volar approach to distal radius fractures. J Hand Surg Am. 2008 Jul-Aug;33(6):958-65. doi: 10.1016/j.jhsa.2008.04.018. PMID 18656773